CLINICAL TRIAL: NCT06374147
Title: "Prapela® SVS Incubator Pad: a Cost-effective Stochastic Vibrotactile Device to Improve the Clinical Course of Infants with Apnea of Prematurity."
Brief Title: "Prapela® SVS Incubator Pad for Apnea of Prematurity
Acronym: Prapela AOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00004467
Record Dates: First submitted 2024-04-16; First posted 2024-04-18 (Actual); Last update posted 2025-03-07 (Actual); Status verified 2025-02

CONDITIONS: Apnea of Prematurity
MeSH Terms: conditions — Apnea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- SVS mattress arm (Experimental): The intervention group will receive standard therapy ( Caffeine Citrate) plus continuous SVS stimulation using the Prapela SVS incubator pad. Treatment with the pad will continue until an infant is apnea-free for 3 days and <2 weeks from anticipated discharge or at the clinician's discretion to discontinue treatment. After ending treatment, clinicians will observe patients 24 hours later and if apnea returns, should re-initiate treatment as needed.
  Interventions: Device: SVS mattress
- Standard (No Intervention): The control group will receive only standard therapy, using an inert pad (identical to the SVS pad, its controller, and green light, but without the transducer and therefore incapable of vibration), in order to mask caregivers

INTERVENTIONS:
Device: SVS mattress — The intervention group will receive standard therapy plus continuous SVS stimulation using the Prapela SVS incubator pad. The control group will receive only standard therapy, using an inert pad (identical to the SVS pad, its controller, and green light, but without the transducer and therefore incapable of vibration), in order to mask caregivers. Treatment with the pad will continue until an infant is apnea-free for 3 days and <2 weeks from anticipated discharge or at the clinician's discretion to discontinue treatment. After ending treatment, clinicians will observe patients 24 hours later and if apnea returns, should re-initiate treatment as needed. At 1 and 2 years of age, parents will be contacted for a brief telephone follow up survey to assess neurological development
  Arms: SVS mattress arm

SUMMARY:
The study proposes to complete the development of and then establish the safety, efficacy, and clinical risk/benefit of a novel hospital incubator pad with stochastic vibrotactile stimulation (SVS) that will provide a complementary treatment and the first improvement in the clinical management of apnea of prematurity (AOP) in over 20 years. Currently, the only approved therapy for AOP is Caffeine Citrate. The SVS mattress pad can prove to be an effective, non-invasive adjunct to Caffeine Citrate for preterm infants with potential to shorten the need for respiratory support as well as overall shortened length of stay.

DETAILED DESCRIPTION:
The study proposes to complete the development of and then establish the safety, efficacy, and clinical risk/benefit of a novel hospital incubator pad that will provide a complementary treatment and the first improvement in the clinical management of apnea of prematurity (AOP) in over 20 years. Defined as cessation of breathing for 20 seconds or longer or a shorter pause accompanied by hypoxemia, AOP is a major morbidity among preterm infants and a significant healthcare burden. AOP affects 70% of all early preterm births (<34 weeks gestational age) and nearly all at ≤ 28 weeks' gestation. In the United States in 2020, the total annual direct costs associated with AOP exceeded $12 billion. While there is no consensus for treating AOP, common interventions include positional techniques, caffeine citrate, manual tactile stimulation, and supplemental oxygen for hypoxemia. Caffeine citrate is the first line of therapy as it decreases apneic episodes and reduces the need for assisted ventilation. At recommended doses, caffeine has been proven safe and effective. However, in the sole trial supporting its FDA clearance, a majority of newborns treated with caffeine citrate continued to experience apnea events. In 2015, a clinical study using a stochastic vibrotactile stimulation (SVS) investigational device reported a 50% reduction in the number of apnea events. Prapela exclusively licensed the SVS technology of the investigational device and has demonstrated technical feasibility replicating the clinically critical stimulation in prototype incubator pads. The broad objective of this SBIR Fast-Track application is to generate the data and documentation necessary for FDA marketing clearance of a novel device to reduce apnea events in preterm newborns. To accomplish this objective, Prapela proposes four Specific Aims: 1) complete development of the SVS incubator pad, 2) demonstrate the safety of the device, 3) determine the clinical efficacy of the SVS incubator pad as an adjunctive therapy to concurrent pharmacological treatment in newborns with AOP, and 4) document the risk/benefit assessment of the device from clinicians caring for AOP patients. Efficacy will be established through a masked, randomized clinical trial with newborns of <33 weeks gestational age, with postmenstrual age (PMA) of <38 weeks at the time of enrollment. The control group will receive standard care only with caffeine citrate and respiratory support and an inert SVS device, while the intervention group will receive standard therapy concurrent with the Prapela SVS device. The primary outcome measure will be the mean number of apnea events in the three days after study entry, with a reduction in apnea events of 30% or more considered clinically significant. Questionnaires administered at the end of each experimental period to the clinicians present on the final shift will capture the risk/benefit assessment. The successful completion of the project will provide the data and documentation necessary for FDA marketing clearance and commercialization of our SVS incubator pad as a purpose-built device to improve clinical outcomes of preterm infants with AOP

ELIGIBILITY:
Inclusion Criteria:

* 22 week 0 days-32 weeks 6 days gestational age (preterm)
* Either sex
* Single birth
* At least 4 clinically documented apnea events in the previous 24 hours
* Caffeine citrate at least 5 mg/kg/day dosing, with or without respiratory support oxygen, nasal cannula, or CPAP without and added rate or pressure support, if considered necessary by the clinical team)

Exclusion Criteria:

* Intubation and mechanical ventilation, or non-invasive positive pressure ventilation (NIPPV) if not intubated, or pressure support breaths while on CPAP.
* Refusal or withdrawal of consent
* Major congenital malformations (not including patent ductus arteriosus, small hernia)
* Known disorder of breathing other than apnea of prematurity (e.g., congenital central hypoventilation syndrome, laryngotracheomalacia)
* Caffeine citrate dosing exceeding FDA recommended dosing in the first 24 hours, if deemed necessary by the clinical team

Ages: 0 Days to 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Estimated)
Dates: Start 2025-02-06 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in apnea rate | 7-28 days of intervention
  The primary outcome is a single continuous measure, the change in (AOP), days 0-12 inclusive, from the baseline apneic rate assessed during the 24-hour run-in period, when all infants are treated on standard CC dosing prior to randomization on day 0.

SECONDARY OUTCOMES:
Secondary Outcome measure | 0 to12 days and 0 to28 days
  Secondary outcome to be assessed 0 to12 days and 0 to 28 days, inclusive:
  - Change in rate of apneic related oxygen desaturation events (SpO2<80 and <90%)
Secondary Outcome measure | 0 to12 days and 0 to28 days
  Secondary outcomes to be assessed 0 to12 days and 0 to 28 days, inclusive:
  - Change in rate of apneic associated bradycardia events (HR < 100beats per/minute)
Secondary Outcome measure | 0 to12 days and 0 to28 days
  Secondary outcomes to be assessed 0 to12 days and 0 to 28 days, inclusive:
  - Cumulative apneic events
Secondary Outcome measures | 0 to12 days and 0 to28 days
  Secondary outcomes to be assessed 0 to12 days and 0 to 28 days, inclusive:
  - Cumulative dosing and length of caffeine citrate treatment

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Alabama, Birmingham, Alabama
  - Tufts Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No